CLINICAL TRIAL: NCT04641481
Title: An Event-Driven, Phase 3, Randomized, Double-blind, Placebo-controlled, Multicenter Study to Evaluate Efficacy, Safety, Immunogenicity, Lot-to-Lot Consistency of BBV152, a Whole-Virion Inactivated SARS-CoV-2 Vaccine in Adults≥18 Yrs of Age
Brief Title: An Efficacy and Safety Clinical Trial of an Investigational COVID-19 Vaccine (BBV152) in Adult Volunteers
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Bharat Biotech International Limited (Industry)
Collaborators: Indian Council of Medical Research (Other Government); Iqvia Pty Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: BBIL/BBV152-C/2020; BBIL/BBV152-C/2020 (Other: Bharat Biotech International Ltd)
Record Dates: First submitted 2020-11-09; First posted 2020-11-23 (Actual); Last update posted 2021-03-19 (Actual); Status verified 2021-03

CONDITIONS: Covid19; SARS-CoV Infection
MeSH Terms: conditions — COVID-19; Severe Acute Respiratory Syndrome | interventions — BBV152 COVID-19 vaccine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: All vaccine and placebo formulations are at a volume of 0.5mL per dose filled into a single-use glass vial. The appearance, color, and viscosity are identical across all vaccine and control formulations.
  Participants, investigators, study coordinators, study-related personnel, and the sponsor will be blinded to the treatment group allocation (excluding an unblinded CRO, who is tasked with the dispatch and labeling of vaccine vials and the generation of the master randomization code). Participants will be assigned a computer-generated randomization code that maintains blinding. The blinded study nurse is responsible for vaccine preparation and administration. Each vial contains a unique code that ensured appropriate blinding.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study vaccine (Experimental): BBV152B (6µg-Algel-IMDG)
  Interventions: Biological: BBV152
- Placebo (Placebo Comparator): Phosphate buffered saline with Alum (without antigen)
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: BBV152 — BBV152 (6µg-Algel - Imidazoquinoline)
  Arms: Study vaccine
Biological: Placebo — Placebo (PBS+Alum, without antigen)
  Arms: Placebo

SUMMARY:
The BBV152 vaccine is being developed to prevent COVID-19, the disease resulting from Severe Acute Respiratory Syndrome coronavirus (SARS-CoV-2) infection. The study is designed to primarily evaluate the efficacy, safety, and immunogenicity of BBV152 to prevent COVID-19 for up to 1 year after the second dose of BBV152.

DETAILED DESCRIPTION:
This is a phase 3 Event-Driven, randomized, double-blind, placebo-controlled, multicentre study to Evaluate the Efficacy, Safety, and Immunogenicity of BBV152, a Whole-Virion Inactivated SARS-CoV-2 Vaccine in Volunteers aged 18 years and above.

A total of 25,800 subjects will be enrolled and randomized in a 1:1 ratio to receive the BBV152 vaccine and control. All participants will be assessed for efficacy and safety endpoints and provide a Nasopharyngeal(NP) swab and blood sample before the first dose of IP. The NP swab and blood collected will be subject to RT-PCR and Anti-SARS-CoV-2 IgG antibodies. The results of this will not affect the enrollment of the participant. Participants who are found to be positive for either RT-PCR Or Anti-SARS-CoV-2 IgG antibodies will be excluded from the primary efficacy analysis. A safety follow-up will be done for all.

In addition, sites will be segregated based on the study objectives:

Category 1 (Symptomatic): In addition to administering the IP, a series of post-dose telephonic follow-up visits will be scheduled to detect suspect symptomatic COVID-19 infections. If a suspect is identified, a nasopharyngeal sample will be collected from the participant for detecting the presence of COVID-19 infection. Telephonic follow-up will occur at 15 Day intervals.

Category 2 (Symptomatic/Asymptomatic): In addition to administering the IP, a series of post-dose Nasopharyngeal samples for detecting an incidence of asymptomatic COVID-19 infection at 1-Month intervals will be collected.

Category 3 (Symptomatic/Asymptomatic+Immunogenicity): In addition to administering the IP and collecting NP samples, a series of blood samples will be collected for analyzing serum for immunological assessments.

The Phase 3 study will follow randomized study participants for efficacy until virologically confirmed (RT-PCR positive) symptomatic COVID-19 participants will be eligible for the primary efficacy analysis. After reaching the target number (n=130) of symptomatic COVID-19 cases, the study will continue to assess safety until the completion of the study duration. It is planned to continue the Phase 3 trial until 130 study participants in the per-protocol population develop PCR-confirmed symptomatic COVID-19 disease during follow-up beginning 14 days after the second dose of vaccine or placebo. We estimate that approximately 25,800 participants should be randomized to accrue these 130 events. The Lot-to-Lot consistency (Immunogenicity) study will be nested within the Phase 3 (Efficacy) study (in three selected sites). The Immunogenicity study will assess the immune response of a 2-dose regimen of BBV152B vaccine through geometric mean titers (GMTs) by neutralizing antibody, S-protein, and RBD specific anti-IgG binding titer in a subset of 600 (450 vaccine: 150 placebo) participants, across three consecutive manufacturing Lots. Data generated through Day 56 (Month 2) will be unblinded only to the biostatistician for evaluation of immune responses in the Immunogenicity subset.

Formal interim analyses are planned when approximately 1/3 and 2/3 of the target number of participants with confirmed symptomatic COVID-19 have been accrued, to determine whether the sample size and/or length of follow-up should be increased. This interim report containing safety and immunogenicity data will be submitted to CDSCO.

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide written informed consent and availability to fulfill the study requirements.
* Participants of either gender of aged 18 years and above.
* Participants with good general health as determined by the discretion of the investigator, or participants with stable medical conditions. A stable medical condition is defined as a disease not requiring significant change in therapy or hospitalization or worsening disease during the 3 months before enrolment.
* For a female participant of child-bearing potential, planning to avoid becoming pregnant (use of an effective method of contraception or abstinence) from the time of study enrolment until at least eight weeks after the last vaccination.
* Male subjects of reproductive potential: Use of condoms to ensure effective contraception with the female partner and to refrain from sperm donation from first vaccination until at least 3 months after the last vaccination.
* Agrees not to participate in another clinical trial at any time during the study period.
* Agrees not to take any COVID-19 licensed vaccination for the entire duration of the study.
* Agrees to remain in the study area for the entire duration of the study.
* Willing to allow storage and future use of biological samples for future research

Exclusion Criteria:

* History of any other COVID-19 investigational or licensed vaccination.
* Known history of SARS-CoV-2 infection, as declared by the subject.
* For women, positive urine pregnancy test before the first dose of vaccination, or any time during the study period.
* Temperature >38.0°C (100.4°F) or symptoms of an acute self-limited illness such as an upper respiratory infection or gastroenteritis within three days prior to each dose of vaccine.
* Resident of COVID-19 infection in the same household.
* Known case of HIV, hepatitis B, or hepatitis C infection.
* Receipt of any licensed/experimental vaccine within four weeks before enrolment in this study.
* Receipt of immunoglobulin or other blood products within the three months before vaccination in this study.
* Immunosuppression as a result of an underlying illness or treatment with immunosuppressive or cytotoxic drugs, or use of anticancer chemotherapy or radiation therapy within the preceding 36 months.
* Immunoglobulins, anti-cytokine antibodies, and blood products within 6 months prior to study vaccination, during, and 21 days following the last dose of vaccination.
* Pregnancy, lactation, or willingness/intention to become pregnant during the first 6 months after enrolment.
* Severe and/or uncontrolled cardiovascular disease, respiratory disease, gastrointestinal disease, liver disease, renal disease, an endocrine disorder, and neurological illness (mild/moderate well-controlled comorbidities are allowed)

Re-Vaccination Exclusion Criteria

* Pregnancy.
* History of virologically (RT-PCR) confirmed SARS-CoV-2 infection
* Anaphylactic reaction following administration of the investigational vaccine.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25800 (Actual)
Dates: Start 2020-11-16 (Actual); Primary Completion 2021-01-08 (Actual); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
First occurrence of Virologically confirmed (RT-PCR positive) symptomatic cases of COVID-19. | Day 42 to Month 12
  (RT-PCR positive) symptomatic cases of COVID-19.

SECONDARY OUTCOMES:
First occurence of Virologically confirmed (RT-PCR positive) symptomatic cases of COVID-19 based on the case definition for the secondary efficacy symptomatic endpoint. | Day 42 to Month 12
  (RT-PCR positive) symptomatic cases of COVID-19.
Virologically confirmed (RT-PCR positive) severe cases of COVID-19 | Day 42 to Month 12
  (RT-PCR positive) severe symptomatic cases of COVID-19.
Virologically confirmed COVID-19 cases of any severity occurring among participants 18 through 59 years of age and ≥60 years of age. | Day 42 to Month 12
  (RT-PCR positive) symptomatic cases of COVID-19
Virologically confirmed COVID-19 asymptomatic and symptomatic cases occurring from two weeks after the second vaccination. | Day 42 to Month 12
  (RT-PCR positive) asymptomatic/symptomatic cases of COVID-19.
Reactogenicity and Safety | Day 42 to Month 12
  Solicited, Unsolicited, Serious Adverse Events
The occurrence of enhanced respiratory disease episodes. | Day 42 to Month 12
  Reported by participant/documented in hospital records throughout the trial.
Immunogenicity: Lot-to-Lot consistency of three consecutive GMP Lots | Day 0 to Day 42
  Assessed based Wild-type SARS-CoV-2 Specific Neutralizing Antibody (nAb)
Geometric Mean Titer (GMT) of SARS-CoV-2 Specific Neutralizing Antibody (nAb) | Day 0 to Month 12
  Specific Neutralizing Antibody (nAb)

CONTACTS AND LOCATIONS:
Overall Officials: Dr Chadramani Singh, Principal Investigator — All India Institute of Medical Sciences; Dr Sanjay Kumar Rai, Principal Investigator — All India Institute of Medical Sciences Delhi; Dr Azhar Ali Khan, Principal Investigator — Baba Raghav Das Medical Gorakhpur; DrAnil Kumar Pandey, Principal Investigator — ESIC Medical College and Hospital Faridabad; Dr Simmi Dube, Principal Investigator — Gandhi Medical College, Bhopal; Dr Anjan Jyoti Talukdar, Principal Investigator — Gauhati Medical College & Hospital Assam; Dr Priti Meshram, Principal Investigator — Grant Government Medical College and Sir J.J. Group of Hospitals Mumbai; Dr Laxmi S Kumari, Principal Investigator — Guntur Medical College ,Guntur; Dr Shiva Narang, Principal Investigator — Guru Teg Bahadur Hospital; Dr E Venkat Rao, Principal Investigator — Institute of Medical Sciences and SUM Hospital Odisha; Dr P Venugopal, Principal Investigator — King George Hospital Visakhapatnam; Dr. N.T. Awad, Principal Investigator — Lokamanya tilak Municipal Medical College and General hospital Mumbai; Dr Pajanivel Ranganadin, Principal Investigator — Mahatma Gandhi Medical College& Research Institute Pondicherry; Dr Prabhakar Reddy, Principal Investigator — Nizam's Institute of Medical Sciences Hyderabad; Dr Raghavendra Gumashta, Principal Investigator — Peoples university Bhopal; Dr Tapan Kumar Saikia, Principal Investigator — Prince Aly Khan Hospital Mumbai; Dr Savita Verma, Principal Investigator — Pt BO Sharma,PGIMS/UHS. Rohtak, Haryana; Dr Manish Multani, Principal Investigator — Rahate Surgical Hospital ,Nagpur; Dr Sagar Vivek Redkar, Principal Investigator — Redkar Hospital and Research Centre Goa; Dr Meghana Murthy, Principal Investigator — Vagus Super speciality hospital,Bangalore; Dr Akshata, Principal Investigator — Vydehi Institute of Medical Sciences and Research Centre,Bangalore; Dr T S Selvavinayagam, Principal Investigator — Directorate of Public Health and Preventive Medicine,Chennai; Dr Suman Kanungo, Principal Investigator — ICMR-National Institute of Cholera and Enteric Diseases,West Bengal; Dr Mohammad Shameem, Principal Investigator — Aligarh Muslim University,Uttar Pradesh; Dr Parul Bhatt, Principal Investigator — Gmers Medical College and Civil Hospital,Ahmedabad
Locations (1):
- Pt BD SHARMA,PGIMS/UHS, Rohtak, Haryana, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ella R, Reddy S, Blackwelder W, Potdar V, Yadav P, Sarangi V, Aileni VK, Kanungo S, Rai S, Reddy P, Verma S, Singh C, Redkar S, Mohapatra S, Pandey A, Ranganadin P, Gumashta R, Multani M, Mohammad S, Bhatt P, Kumari L, Sapkal G, Gupta N, Abraham P, Panda S, Prasad S, Bhargava B, Ella K, Vadrevu KM; COVAXIN Study Group. Efficacy, safety, and lot-to-lot immunogenicity of an inactivated SARS-CoV-2 vaccine (BBV152): interim results of a randomised, double-blind, controlled, phase 3 trial. Lancet. 2021 Dec 11;398(10317):2173-2184. doi: 10.1016/S0140-6736(21)02000-6. Epub 2021 Nov 11. PMID 34774196